CLINICAL TRIAL: NCT03481543
Title: Effectiveness of Bronchodilator Nebulization With and Without Noninvasive Ventilation During Respiratory Failure in Chronic Obstructive Pulmonary Disease
Brief Title: Effectiveness of Bronchodilator Nebulization With and Without Noninvasive Ventilation in COPD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: National University Health System, Singapore (Other)
Responsible Party: Principal Investigator, Amartya Mukhopadhyay, Principal investigator, National University Health System, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSRB 2017/00990
Record Dates: First submitted 2018-03-15; First posted 2018-03-29 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Type 2 Respiratory Failure
Keywords: Chronic Obstructive Pulmonary Disease (COPD); Nebulization; Respiratory failure; Non-invasive ventilation(NIV)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoventilation; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-line nebulization through NIV mask (Experimental): Bronchodilator nebulization is given through NIV circuit.
  Interventions: Procedure: In-line nebulization through NIV mask
- Off-NIV nebulization (Active Comparator): Bronchodilator nebulization is given during which NIV mask is taken off for a short time and reapplied when nebulization is finished.
  Interventions: Procedure: Off-NIV nebulization

INTERVENTIONS:
Procedure: In-line nebulization through NIV mask — In-line nebulization will be given through NIV circuit.
  Arms: In-line nebulization through NIV mask
Procedure: Off-NIV nebulization — Bronchodilator nebulization is given during which NIV mask is taken off for a short time and reapplied when nebulization is finished..
  Arms: Off-NIV nebulization

SUMMARY:
The study aim to evaluate effectiveness of two bronchodilator nebulization strategies in patients with acute decompensated type 2 respiratory failure due to acute exacerbation of chronic obstructive pulmonary disease..

DETAILED DESCRIPTION:
Decompensated type 2 respiratory failure during acute exacerbation of chronic obstructive pulmonary disease (COPD) is treated with non-invasive ventilation (NIV) and nebulized bronchodilators. Nebulization during NIV can be applied by two methods: in-line nebulization through NIV mask and off-NIV nebulization during which NIV mask is taken off for a short time and reapplied when nebulization is finished.

This study is a prospective randomized controlled trial to compare in-line nebulization through NIV versus off- NIV nebulization. After starting NIV in eligible COPD patients with type 2 respiratory failure, the baseline end-expiratory lung impedance (EELI) will be measured. Patient is randomized to receive either in-line or off-NIV nebulization. EELI will be measured again following completion of the nebulization, 15min after NIV is restarted (off-NIV group) or continued (in-line group). Ultrasound measurement of the thickness of the diaphragm will be recorded at baseline, 15min after NIV is restarted (off-NIV group) or continued (in-line group) and 48 hours after stopping the NIV. The main outcome measure, difference in mean end expiratory lung volume at 15min after NIV is restarted (off-NIV group) or continued (in-line group) between the two nebulization methods will be compared using independent sample T test. Thickness of the diaphragm and changes in the arterial blood gases (in terms of pH and carbon-di-oxide) will be compared between in-line nebulization and off-NIV nebulization.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥21 years.
2. Known or suspected COPD (defined by a ratio of Forced Expiratory Volume in 1 second (FEV1) to Forced Vital Capacity (FVC) of less than 0.7).
3. Acute decompensated type 2 respiratory failure (ABG pH ≤ 7.35 and PaCO2>45mmHg).
4. Clinical decision made to start NIV.

Exclusion Criteria:

1. Other acute decompensated type 2 respiratory failure related conditions (e.g. neuromuscular, heart failure etc.).
2. Pneumonia present in the chest radiograph.
3. Other conditions which may change lung impedance (e.g. heart failure or lung fibrosis).

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Difference in mean end-expiratory lung volumes between the two nebulization methods. | At baseline (approximately 15min after starting NIV) to approximately 15min after restarting (or continuing NIV) following the nebulization.
  End-expiratory lung volumes between in-line nebulization and off-NIV nebulization.

SECONDARY OUTCOMES:
Thickness of the diaphragm (by ultrasound) between in-line nebulization and off-NIV nebulization. | At baseline (approximately 15min after starting NIV) to approximately 15min after restarting (or continuing NIV) following the nebulization and repeated 48hours after stopping NIV.
  Measure thickness of the diaphragm between inspiration and expiration.
Changes in arterial blood gases in terms of pH and carbon dioxide between in-line. nebulization and off-NIV nebulization. | At baseline (approximately 15min after starting NIV) to approximately 15min after restarting (or continuing NIV) following the nebulization.
  Measure changes of arterial blood gases between in-line nebulization and off-NIV. nebulization. Differences in pH (absolute,no unit) and carbon dioxide (in mmHg) will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Amartya Mukhopadhyay, MBBS, Principal Investigator — National University Health System
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brochard L, Mancebo J, Wysocki M, Lofaso F, Conti G, Rauss A, Simonneau G, Benito S, Gasparetto A, Lemaire F, et al. Noninvasive ventilation for acute exacerbations of chronic obstructive pulmonary disease. N Engl J Med. 1995 Sep 28;333(13):817-22. doi: 10.1056/NEJM199509283331301. PMID 7651472
- [Result] Vivier E, Mekontso Dessap A, Dimassi S, Vargas F, Lyazidi A, Thille AW, Brochard L. Diaphragm ultrasonography to estimate the work of breathing during non-invasive ventilation. Intensive Care Med. 2012 May;38(5):796-803. doi: 10.1007/s00134-012-2547-7. Epub 2012 Apr 5. PMID 22476448
- [Result] Pauwels RA, Buist AS, Calverley PM, Jenkins CR, Hurd SS; GOLD Scientific Committee. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease. NHLBI/WHO Global Initiative for Chronic Obstructive Lung Disease (GOLD) Workshop summary. Am J Respir Crit Care Med. 2001 Apr;163(5):1256-76. doi: 10.1164/ajrccm.163.5.2101039. No abstract available. PMID 11316667